CLINICAL TRIAL: NCT03601988
Title: A Randomized Phase III Trial of Postoperative Chemotherapy or Chemo-radiotherapy for Locally Advanced Gastric Cancer After D2 Resection
Brief Title: Phase III Trial of Adjuvant Chemo-radiotherapy After D2 Surgery of Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Head of the cancer center, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJCC007
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; radiotherapy; postoperative
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: All patients randomized to receive chemotherapy or chemo-radiotherapy after D2 surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator): Adjuvant chemotherapy group receive 8 cycles of XELOX (Oxaliplatin 130mg/m2, ivdrip, D1,capecitabine 1000mg po, Bid, D1-14, Q21D)
  Interventions: Drug: Chemotherapy
- Chemo-radiotherapy (Experimental): Adjuvant chemo-radiotherapy group receive 6 cycles of XELOX (Oxaliplatin 130mg/m2, ivdrip, D1, capecitabine 1000mg po, Bid, D1-14, Q21D) and concurrent chemo-radiotherapy (capecitabine 825mg po, Bid, d1-5, QW)
  Interventions: Radiation: Concurrent chemo-radiotherapy

INTERVENTIONS:
Radiation: Concurrent chemo-radiotherapy — Experimental group receive 6 cycles of XELOX chemotherapy and concurrent chemo-radiotherapy. The radiotherapy dose of 45Gy in 25 fractions delivered by IMRT Radiotherapy
  Arms: Chemo-radiotherapy
Drug: Chemotherapy — Chemotherapy group receive 8 cycles of XELOX.
  Arms: Chemotherapy

SUMMARY:
The purpose of this study is to explore the efficacy of adjuvant radiotherapy for D2 resected gastric cancer

DETAILED DESCRIPTION:
The radiotherapy dose of 45Gy in 25 fractions as adjuvant treatment after D2 surgery for gastric cancer

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75；
2. Had histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction；
3. ECOG 0-1；
4. Subjects has to voluntarily join the study and sign the Informed Consent Form for the study;
5. D2 and R0 resection;
6. Locally advanced (UICC stage, T4, N2, N3) gastric cancer after surgery;
7. More than 15 lymph nodes;
8. Adequate organ function as defined below: Hematologic ANC ≥ 2*109/L, Platelets ≥ 100*109/L, AST and ALT ≤ 2.5×ULN, TBIL ≤ 1.5×ULN.

Exclusion Criteria:

1. Previous radiotherapy or chemotherapy；
2. Inadequate organ function;
3. Pregnant or lactating women or women of childbearing potential.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2018-07-28 (Estimated); Primary Completion 2020-07-28 (Estimated); Study Completion 2022-07-28 (Estimated)

PRIMARY OUTCOMES:
DFS | 36 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months

SECONDARY OUTCOMES:
OS | 36 months
  From date of randomization until the date of first documented death from any cause, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, MD,PhD, Study Chair — Tongji Hospital
Locations (1):
- Tongji hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park SH, Sohn TS, Lee J, Lim DH, Hong ME, Kim KM, Sohn I, Jung SH, Choi MG, Lee JH, Bae JM, Kim S, Kim ST, Park JO, Park YS, Lim HY, Kang WK. Phase III Trial to Compare Adjuvant Chemotherapy With Capecitabine and Cisplatin Versus Concurrent Chemoradiotherapy in Gastric Cancer: Final Report of the Adjuvant Chemoradiotherapy in Stomach Tumors Trial, Including Survival and Subset Analyses. J Clin Oncol. 2015 Oct 1;33(28):3130-6. doi: 10.1200/JCO.2014.58.3930. Epub 2015 Jan 5. PMID 25559811
- [Background] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Background] Noh SH, Park SR, Yang HK, Chung HC, Chung IJ, Kim SW, Kim HH, Choi JH, Kim HK, Yu W, Lee JI, Shin DB, Ji J, Chen JS, Lim Y, Ha S, Bang YJ; CLASSIC trial investigators. Adjuvant capecitabine plus oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): 5-year follow-up of an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1389-96. doi: 10.1016/S1470-2045(14)70473-5. Epub 2014 Oct 15. PMID 25439693
- [Background] Macdonald JS, Smalley SR, Benedetti J, Hundahl SA, Estes NC, Stemmermann GN, Haller DG, Ajani JA, Gunderson LL, Jessup JM, Martenson JA. Chemoradiotherapy after surgery compared with surgery alone for adenocarcinoma of the stomach or gastroesophageal junction. N Engl J Med. 2001 Sep 6;345(10):725-30. doi: 10.1056/NEJMoa010187. PMID 11547741
- [Background] Kim Y, Park SH, Kim KM, Choi MG, Lee JH, Sohn TS, Bae JM, Kim S, Lee SJ, Kim ST, Lee J, Park JO, Park YS, Lim HY, Kang WK. The Influence of Metastatic Lymph Node Ratio on the Treatment Outcomes in the Adjuvant Chemoradiotherapy in Stomach Tumors (ARTIST) Trial: A Phase III Trial. J Gastric Cancer. 2016 Jun;16(2):105-10. doi: 10.5230/jgc.2016.16.2.105. Epub 2016 Jun 24. PMID 27433396
- [Background] Lee J, Lim DH, Kim S, Park SH, Park JO, Park YS, Lim HY, Choi MG, Sohn TS, Noh JH, Bae JM, Ahn YC, Sohn I, Jung SH, Park CK, Kim KM, Kang WK. Phase III trial comparing capecitabine plus cisplatin versus capecitabine plus cisplatin with concurrent capecitabine radiotherapy in completely resected gastric cancer with D2 lymph node dissection: the ARTIST trial. J Clin Oncol. 2012 Jan 20;30(3):268-73. doi: 10.1200/JCO.2011.39.1953. Epub 2011 Dec 19. PMID 22184384